CLINICAL TRIAL: NCT04469712
Title: Long-term Outcomes of Bariatric Patients Treated With Gastric Bypass or Single-anastomosis Sleeve Ileal Bypass (SASI Bipartition)
Brief Title: Non-randomized Prospective Comparison Between SASI Bipartition and RYGB
Status: Active, not recruiting | Type: Observational
Sponsor: Aleris Hospital (Other)
Responsible Party: Principal Investigator, Ebrahim Aghajani, Gastrointestinal Surgeon, PhD, Principal investigator, Aleris Hospital
Other Study IDs: 66095
Record Dates: First submitted 2020-07-03; First posted 2020-07-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Morbid; Metabolic Syndrome; Bariatric Surgery Candidate; Postoperative Complications
Keywords: Gastric Bypass,; SASI Bipartition; Weight loss; GERD; Internal Hernia
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Postoperative Complications; Weight Loss; Gastroesophageal Reflux; Internal Hernia | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SASI Bipartition: Subjects submitted to SASI Bipartition
  Interventions: Procedure: SASI Bipartition
- Roux-en-Y gastric bypass: Subjects submitted to gastric bypass
  Interventions: Procedure: Gastric bypass

INTERVENTIONS:
Procedure: SASI Bipartition — SASI Bipartition is performed with a sleeve gastrectomy over a 32 French gastric bougie and a 300 cm common limb. Side-to-side gastroileostomy with a diameter of approximately 2.5 cm at the anterior part of antrum, 6 cm proximal to pylorus.
  Other Names: Single-anastomosis Sleeve Ileal Bypass
  Groups: SASI Bipartition
Procedure: Gastric bypass — A small gastric pouch (15 mL) is created, and the jejunum brought up as an antecolic and antegastric fashion. Routine limb lengths were 150 cm for the alimentary limb and 60 cm for the bilio-pancreatic limb. Both mesenteric defects are closed with the Endohernia® stapler.
  Other Names: Roux-en-Y gastric bypass
  Groups: Roux-en-Y gastric bypass

SUMMARY:
The main aim of this project is to assess the safety and efficiency of the SASI Bipartition.

DETAILED DESCRIPTION:
The Roux-en-Y Gastric Bypass (RYGB) is the procedure of choice in morbid obesity with metabolic disorders in most of the reference centers. Recent data describes the SASI Bipartition as being as efficient on weight loss and co-morbidities as the RYGB, with the advantage of being less technically difficult and less morbidity. In order to draw definite conclusions regarding the procedure, larger series with longer follow-up are necessary.

Patients with BMI over 40, or with BMI over 35 with comorbidities are offered SASI Bipartition with 300 cm common limb or standard RYGB. Follow up is performed through visits at 3, 12, 24, 36, 48, and 60 months after surgery.

Results on weight loss, comorbidities resolution, complications, and need of supplements are registered.

ELIGIBILITY:
Inclusion Criteria:

- Morbid obesity with BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 associated with one or more co-morbidities (type 2 diabetes, arterial hypertension, sleep apnea, dyslipidemia, arthritis)

Exclusion Criteria:

* Mental diseases
* Drug addiction
* Alcoholic
* Malignancy
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients approved for bariatric surgery at Bariatric Clinic, Aleris Hospital, Norway
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Weight change | 3 to 60 months after surgery
  Measured as percent of Excess Weight Loss (%EWL) using the following formula:
  ((weight at each study visit - initial weight) / (initial weight - ideal weight)) X 100
Waist size change | 3 to 60 months after surgery
  Waist size (in cm)
Medical and surgical complication | 3 to 60 months after surgery
  According to Clavien-Dindo classification
Operative time | During surgery
  Expressed in minutes
Hemoglobin | before surgery up to 60 months after surgery
  Measurement of Hemoglobin will explore the nutritional status of patients. Results will be expressed in g/l
Albumin | before surgery up to 60 months after surgery
  Measurement of albumin will explore the nutritional status of patients. Results will be expressed in g/l
Ferritin | before surgery up to 60 months after surgery
  Measurement of ferritin will explore the nutritional status of patients. Results will be expressed in microg/l
Iron | before surgery up to 60 months after surgery
  Measurement of iron will explore the nutritional status of patients. Results will be expressed in micromol/l
Parathyroid hormone (PTH) | before surgery up to 60 months after surgery
  Measurement of PTH will explore the nutritional status of patients. Results will be expressed in pmol/L
Vitamin B12 | before surgery up to 60 months after surgery
  Measurement of vitamin B12 will explore the nutritional status of patients. Results will be expressed in pmol/l
Vitamin D | before surgery up to 60 months after surgery
  Measurement of vitamin D will explore the nutritional status of patients. Results will be expressed in nmol/l

SECONDARY OUTCOMES:
Fasting glycemia | before surgery up to 60 months after surgery
  Measurement of fasting glycemia will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
HbA1c | before surgery up to 60 months after surgery
  Measurement of HbA1c will explore the Metabolic efficiency of surgery. Results will be expressed in %
Triglycerides | before surgery up to 60 months after surgery
  Measurement of triglycerides will explore the Metabolic of surgery. Results will be expressed in mmol/l
Cholesterol | before surgery up to 60 months after surgery
  Measurement of cholesterol will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
HDL | before surgery up to 60 months after surgery
  Measurement of HDL will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
LDL | before surgery up to 60 months after surgery
  Measurement of LDL will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
Antidiabetic drugs | 3 to 60 months after surgery
  Evolution of antidiabetic drugs will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Antilipidemic drugs | 3 to 60 months after surgery
  Evolution of antilipidemic drugs will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Antihypertensive drugs | 3 to 60 months after surgery
  Evolution of antihypertensive drugs will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Use of Continuous Positive Airway Pressure for Obstructive Sleep Apnea (OSA) | 3 to 60 months after surgery
  Evolution of the use of Continuous Positive Airway Pressure will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of persistence or not of OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Aghajani, PhD, Principal Investigator — Aleris Hospital
Locations (1):
- Aleris Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
The results of the study will be published in a scientific journal.

REFERENCES:
- [Background] Aghajani E, Nergaard BJ, Leifson BG, Hedenbro J, Gislason H. The mesenteric defects in laparoscopic Roux-en-Y gastric bypass: 5 years follow-up of non-closure versus closure using the stapler technique. Surg Endosc. 2017 Sep;31(9):3743-3748. doi: 10.1007/s00464-017-5415-2. Epub 2017 Feb 15. PMID 28205037
- [Background] Santoro S, Castro LC, Velhote MC, Malzoni CE, Klajner S, Castro LP, Lacombe A, Santo MA. Sleeve gastrectomy with transit bipartition: a potent intervention for metabolic syndrome and obesity. Ann Surg. 2012 Jul;256(1):104-10. doi: 10.1097/SLA.0b013e31825370c0. PMID 22609843
- [Background] Mahdy T, Al Wahedi A, Schou C. Efficacy of single anastomosis sleeve ileal (SASI) bypass for type-2 diabetic morbid obese patients: Gastric bipartition, a novel metabolic surgery procedure: A retrospective cohort study. Int J Surg. 2016 Oct;34:28-34. doi: 10.1016/j.ijsu.2016.08.018. Epub 2016 Aug 19. PMID 27545956
- [Background] Mui WL, Lee DW, Lam KK. Laparoscopic sleeve gastrectomy with loop bipartition: A novel metabolic operation in treating obese type II diabetes mellitus. Int J Surg Case Rep. 2014;5(2):56-8. doi: 10.1016/j.ijscr.2013.12.002. Epub 2013 Dec 10. PMID 24441436
- [Background] Shah K, Johnny Nergard B, Stray Frazier K, Geir Leifsson B, Aghajani E, Gislason H. Long-term effects of laparoscopic Roux-en-Y gastric bypass on metabolic syndrome in patients with morbid obesity. Surg Obes Relat Dis. 2016 Sep-Oct;12(8):1449-1456. doi: 10.1016/j.soard.2016.03.017. Epub 2016 Mar 19. PMID 27387692